CLINICAL TRIAL: NCT04033172
Title: Pyrotinib Plus Fulvestrant in Patients HR+/HER2+ Metastatic Breast Cancer : a Prospective, Single-arm, Single-center Study
Brief Title: Pyrotinib Plus Fulvestrant in Patients With HR+/HER2+ Metastatic Breast Cancer (Pyrotinib+Fulvestrant )
Acronym: Pyrotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2018M-042
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: Metastatic Breast Cancer, Pyrotinib, Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib plus Fulvestrant (Experimental)
  Interventions: Drug: Pyrotinib Plus Fulvestrant

INTERVENTIONS:
Drug: Pyrotinib Plus Fulvestrant — Pyrotinib: 400 mg/d, q.d., p.o. A course of treatment need 28 days. Fulvestrant: 500 mg/m2 q.d. i.m. A course of treatment need 28 day. First course needs extra dose of fulvestrant 500 mg/m2 q.d. i.m. on day 15.

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both HER1, HER2 and HER4 receptors. This study is a single-arm, prospective, single-center clinical study of pyrotinib plus fulvestrant as the therapy HR+/HER2+ metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-75 years old; HR positive and HER2 positive (immunohistochemistry or FISH test confirmed).
2. ECOG score ≤ 2, expected survival ≥ 3 months.
3. Histology or cytology confirmed as breast cancer.
4. Prior to trastuzumab and endocrine therapy and progression/recurrence.
5. At least one RECIST 1.1 defined measurable lesions.
6. Normal function of major organs.

Exclusion Criteria:

1. pregnant or lactating women
2. Patients who have relapsed or progressed within 12 months of end of adjuvant or neoadjuvant therapy, including chemotherapy, target therapy (eg lapatinib， trastuzumab), or other anti-tumor therapy. Except for endocrine therapy.
3. Severe chronic gastrointestinal diseases with diarrhea as the main symptom (such as Crohn's disease, malabsorption, or ≥2 grade diarrhea caused by any cause at baseline).
4. Rapid progress of organ invasion (such as liver and lung disease greater than 1/2 organ area or liver dysfunction, etc.)
5. Patients with central nervous system disorders or mental disorders
6. Bone metastasis lesions only, no other measurable lesions.
7. Hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 100 mmHg) without ideal control.
8. Uncontrolled heart disease.
9. Have congenital long or short QT syndrome or have a family history or personal history of Brugada syndrome.
10. Uncontrolled rain metastasis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Estimated up to 1 year
  Defined as the time from the date of informed consent to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
OS (overall survival) | Estimated up to 1 year
  Defined as the time from the date of informed consent until to the date of death, regardless of the cause of death.
Objective Response Rate (ORR) | Estimated up to 1 year
  Defined as proportion of complete response and partial response according to RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Jian Yue, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No